CLINICAL TRIAL: NCT04581772
Title: A Phase 1 Open-Label, Randomized, Crossover Study to Evaluate the Bioavailability, Effect of Food, Palatability, and Safety of Various DNL343 Oral Formulations in Healthy Participants
Brief Title: A Study to Evaluate the Bioavailability and Safety of DNL343 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-F-0002
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental)
  Interventions: Drug: DNL343; Drug: Placebo
- Cohort B (Experimental)
  Interventions: Drug: DNL343; Drug: Placebo
- Cohort C (Experimental)
  Interventions: Drug: DNL343

INTERVENTIONS:
Drug: DNL343 — Multiple oral doses
  Arms: Cohort A; Cohort B
Drug: Placebo — Single oral dose
  Arms: Cohort A; Cohort B
Drug: DNL343 — Single oral dose
  Arms: Cohort C

SUMMARY:
This is a Phase 1 relative bioavailability study carried out in approximately 24 healthy male subjects and healthy female subjects of non childbearing potential to investigate the effects of formulation and food on the safety, tolerability, and pharmacokinetics (PK) of DNL343.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) ≥18.5 to < 30 kg/m2 and body weight of at least 50 kg
* For women: Must have been surgically sterilized or be postmenopausal.

Key Exclusion Criteria:

* History of clinically significant endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematologic, immunologic, or allergic disease, or other major disorders
* History of malignancy, except fully resected basal cell carcinoma
* History of clinically significant neurologic or psychiatric diseases; head trauma with loss of consciousness; or clinically significant depression or suicidal ideation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
PK parameter: Maximum observed concentration (Cmax) of DNL343 in plasma | Up to 15 days
PK parameter: Time to maximum observed concentration (Tmax) of DNL343 in plasma | Up to 15 days
PK Parameter: Area under the concentration-time curve from time zero to the last quantifiable time point (AUC0-t) of DNL343 in plasma | Up to 15 days
PK parameter: The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL343 in plasma | Up to 15 days

SECONDARY OUTCOMES:
PK parameter: Maximum observed concentration (Cmax) of DNL343 in plasma in the fed versus fasted states | Up to 15 days
PK parameter: Time to maximum observed concentration (Tmax) of DNL343 in plasma in the fed versus fasted states | Up to 15 days
PK Parameter: Area under the concentration-time curve from time zero to the last quantifiable time point (AUC0-t) of DNL343 in plasma in the fed versus fasted states | Up to 15 days
PK parameter: The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL343 in plasma in the fed versus fasted states | Up to 15 days
Incidence of treatment-emergent adverse events (TEAEs) | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsai, MD, Study Director — Denali Therapeutics Inc.
Locations (1):
- Auckland Clinical Studies Ltd., Grafton, Auckland, New Zealand